CLINICAL TRIAL: NCT06978608
Title: Ultrasound and Somatosensory Evaluation of the Median Nerve at the Carpal Canal in Patients With CRPS Type I and Clinical Correlation: Definition of Morphologic Patterns
Brief Title: Ultrasound and Somatosensory Median Nerve Evaluation in CRPS I
Acronym: MEDICUS
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Other Study IDs: Prot.: 0003733 del 2025; Rif CEAVC 28194 (Registry Identifier: Comitato Etico USL Toscana Centro)
Record Dates: First submitted 2025-04-23; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: CRPS (Complex Regional Pain Syndrome) Type I
Keywords: CRPS; MEDIAN NERVE; CARPAL TUNNEL; SENSORY; ULTRASOUND; SOMATOSENSORY
MeSH Terms: conditions — Complex Regional Pain Syndromes; Median Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Budapest Criteria positive for CRPS type I, older than 18 years old: Any specific symptoms will be recorded. Patients will undergo ultrasound examination to analyze on both the healthy and diseased side the morphological aspect of the median nerve at the carpal tunnel level, to address gliding in terms of mm, adhesion between the transverse ligament and flexor tendons. The aim will be to try to define specific predictive morphological patterns relative to the clinical appearance. Sensory nerve conduction velocity (SNCV) of the median-nerve will be evaluated to analyze the somatosensory part of the median nerve and understand the potential use of this as a diagnostic tool.

SUMMARY:
Complex regional pain syndrome (CRPS) is a disorder falling within the sphere of neuropathic pain, characterised by a plethora of symptoms. Regional pain out of proportion to the triggering event is the main presentation, accompanied by allodynia, dysesthesia, thermal asymmetry, trophic changes, oedema and stiffness. Recently, preliminary observational studies have found that the management of patients with CRPS, refractory to pharmacological treatment, by carpal tunnel release may be resolving; This suggests that an irritative carpal tunnel syndrome may be masked as CRPS due to non-specific symptoms and negative electrodiagnostic studies (electromyography-EMG). Classical carpal tunnel syndrome (CTS) is a well-defined clinical condition that can be ascertained by EMG. In contrast, irritative carpal tunnel syndrome has symptoms attributable to CRPS with negative EMG that arises after trauma that required surgery or immobilisation. It is unclear how to define the presence of irritative carpal tunnel syndrome in patients diagnosed as CRPS, and thus how to make a correct diagnosis. Nor is the management of these patients defined. The aim of the research is to analyse all patients with typical symptoms for CRPS to investigate the morphological appearance of the median nerve at the level of the carpal tunnel by means of dynamic ultrasound in comparison with the healthy limb. In addition, in order to quantify the function of the median nerve, investigators will analyse patients by means of a sensory conduction velocity study (SNVC), as common EMG examinations are negative in these patients, while it is possible that the quantification of the sensory part of the nerve may be impaired. In addition, the autonomic component will be investigated by studying the Skin Sudomotor Response (SSR).The hypothesis is that some patients, after an injury that required surgery or immobilisation, develop fibrous soft tissue scarring that creates a kind of space-occupying lesion that compresses the median nerve at the level of the carpal tunnel and reduces its sliding under the transverse ligament of the carpus, a structure that is not elastic and therefore unable to adapt to the volumetric increases within it. The other hypothesis is that the fibrosis and post-traumatic oedema, which is structured, directly involves the median nerve sheath, resulting in irritation. Classical CTS develops due to mechanical trauma, high pressure and ischaemic damage affecting the median nerve and develops as a clinical condition of pure nerve suffering, with symptoms referable to a sensory and motor deficit. In CRPS, on the other hand, allodynia, hyperalgesia, sudomotor and vasomotor abnormalities and trophic changes are all symptoms that may be related, but are not specific, to nerve suffering.

DETAILED DESCRIPTION:
This is a prospective, single-centre, non-profit observational study. The study will be carried out as follows: Patients will be recruited on the presence of positive Budapest Criteria for CRPS type I. Patients suffering from CRPS type I at the SOD of Surgery and Reconstructive Microsurgery of the Hand of the AOU Careggi of Florence (IT) will be included, aged 18 years or older. In particular, each patient will undergo dynamic bilateral wrist ultrasound and the following parameters will be recorded: median nerve sliding in terms of mm, morphological appearance of the median nerve in terms of hypertrophy/hypotrophy, hourglass lesions and relationship with adjacent soft tissues. The surrounding soft tissues will be examined, in particular the tendinous structures within the carpal canal to assess the presence of fibrosis, synovitis and degree of sliding in mm. The ultrasound examination will be performed in all patients with symptoms attributable to CRPS type I. Each patient will also undergo a Neuronographic examination recording the following parameters: Motor conduction velocity (VCM), distal latency of the M response, Sensory Conduction Speed (VCS), amplitude of the sensory action potential (SAP), latency of the sympathetic cutaneous response (SSR) and the following parameters will be recorded: Ultrasound examination will be performed.

The participation of each participant in the study will be superimposed on the performance of the ultrasound and neuronographic examination; 50 patients will be enrolled at this hospital; the study will be conducted exclusively in the Careggi University Hospital. Each patient will be analysed by ultrasound and Neuronographic examination on both healthy and diseased side defining the morphological criteria and Neuronographic parameters of the median nerve based on the findings. The aim will be to try to define specific predictive morphological patterns.

Each patient will continue to be treated both diagnostically and therapeutically, as well as post-therapy monitoring, according to normal clinical practice.

Inclusion criteria

1. patients with a diagnosis of CRPS evaluated at the SOD of Hand Surgery and Reconstructive Microsurgery of the AOUC, Florence (IT)
2. Patients aged 18 years or older
3. Signature of informed consent to participation in the study and processing of related data

Exclusion criteria

1. patients with CRPS type II and therefore with known peripheral nerve injury
2. Patients under 18 years of age

Patients' clinical data (age, sex, treatment provided, clinical outcome) will be extracted from the medical records. Patients will be evaluated periodically on an outpatient basis according to the normal follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with CRPS assessed at the AOUC's Hand Surgery and Reconstructive Microsurgery SOD
2. Patients aged 18 years and over
3. Signature of informed consent for participation in the study and processing of related data

Exclusion Criteria:

1. patients suffering from CRPS type II and therefore with known peripheral nerve injury
2. Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be enrolled at the primary care clinic of the hospital, diagnosed as CRPS type I.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Number of patients with altered gliding and/or presence of adhesion between the median nerve and the flexor tendons and/or transverse carpal ligament in patients affected by CRPS type I | Up to 12 months. From date of recruitment until the date of clinical improvement, assessed up to 12 months
  Ultrasound examination will be done either to the affected and the contralateral side. The median nerve will be studied in terms of gliding of the nerve , adhesions with the flexor tendons and / or the transverse carpal ligament. The presence of hypertrophy will be addressed by measuring the median nerve thickness.

SECONDARY OUTCOMES:
Number of patients with altered sensory nerve conduction velocity study in patients affected by CRPS type I | Up to 12 months. From date of recruitment until the date of clinical improvement, assessed up to 12 months
  Patients that provide a reduction of the velocity at the sensory nerve conduction study as a result of median nerve irritation that manifests as suffering of its somatosensory part.

IPD SHARING:
Plan to Share IPD: No